CLINICAL TRIAL: NCT06070961
Title: Prospective Biological Study to Evaluate the Persistence of COVID-19 Vaccine and Other Vaccines'-Induced Immune Responses in Follicular Lymphoma Patients Undergoing Frontline Induction Immuno-chemotherapy and Anti-CD20 Maintenance
Acronym: FIL_FollVax22
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_FollVax 22
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Follicular Lymphoma
Keywords: Lymphoma; Follicular; Immunochemotherapy; FL; Vaccine; COVID19; SARS-COV-2; Tetanus; Zoster; VZV; Rituximab; obinotuzumab; FOLL19; FIL_FOLL19; diphtheria; Maintenance; Humoral; Cellular; Immunity; Induction
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma; COVID-19; Tetanus; Herpes Zoster; Diphtheria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient affected by advanced Follicular Lymphoma undergoing front-line immunochemotherapy and antiCD-20 maintenance in the FIL_FOLL19 trial
  Interventions: Diagnostic Test: Cellular immunity vs SARS-CoV-2; Diagnostic Test: Humoral immunity vs SARS-CoV-2; Diagnostic Test: Cellular immunity vs Varicella Zoster Virus; Diagnostic Test: Humoral immunity vs Varicella Zoster Virus; Diagnostic Test: Diphtheria toxin-binding IgG; Diagnostic Test: Tetanus toxoid-binding IgG; Diagnostic Test: T-cell populations and markers characterization

INTERVENTIONS:
Diagnostic Test: Cellular immunity vs SARS-CoV-2 — Evaluation of cellular immunity vs SARS-CoV-2 by ELISpot assay
Diagnostic Test: Humoral immunity vs SARS-CoV-2 — Evaluation of Humoral immunity vs SARS-CoV-2 by ELISA assay (IgG anti-RBD and anti-N)
Diagnostic Test: Cellular immunity vs Varicella Zoster Virus — Evaluation of cellular immunity vs VZV by Enzyme-Linked immunoSPOT (ELISPOT) assay
Diagnostic Test: Humoral immunity vs Varicella Zoster Virus — Evaluation of humoral immunity vs VZV by ELISA (VZV gE-binding IgG)
Diagnostic Test: Diphtheria toxin-binding IgG — Evaluation of diphtheria toxin-binding IgG by ELISA assay
Diagnostic Test: Tetanus toxoid-binding IgG — Evaluation of tetanus toxoid-binding IgG by ELISA assay
Diagnostic Test: T-cell populations and markers characterization — Characterization of T-cell populations and markers by flow cytometry

SUMMARY:
This is a prospective biological study evaluating the persistence of COVID-19 vaccine and other vaccines' (zoster, diphtheria and tetanus)-induced immunity in a subgroup patient affected by Follicular Lymphoma requiring treatment undergoing frontline induction immuno-chemotherapy and anti-CD20 maintenance within the prospective FIL_FOLL19 study (NCT05058404).

Blood samples from patients will be collected before and at planned timepoints during treatment to evaluate humoral and cellular immunity against SARS-COV-2, VZV, tetanus and diphtheria and T-cell markers characterization.

DETAILED DESCRIPTION:
Patients (pts) with follicular lymphoma (FL) were reported to be at high risk for hospitalization and death from COVID-19 infection, especially if exposed to anti-CD20 monoclonal antibodies (mAbs)-based therapy. A large amount of studies unequivocally demonstrated that anti-CD20 mAbs-containing therapies typically impair the development of protective levels of neutralizing anti-spike antibodies after immunization with full course of approved mRNA-based COVID-19 vaccines (up to 12 months after last anti-CD20 infusion). Moreover, booster doses seem to induce seroconversion only in a minority of such pts. On the contrary, preliminary findings seem to suggest that a substantial proportion of vaccinated pts with B-cell lymphoma (B-NHL) mount detectable SARS-CoV-2-specific T-cell responses (as measured by assays evaluating IFN-Y secretion after stimulation with SARS-CoV-2 peptides), independently from humoral response status.

For newly diagnosed FL pts current guidelines suggest to complete the vaccination with booster dose(s) before treatment initiation, as anti-CD20 mAbs seems to spare pre-established humoral immunity to COVID-19 vaccine, although data supporting this finding are scanty.5 Furthermore, data about long term persistence of pre-established cellular immunity in this setting are lacking, although preliminary findings in unselected immunosuppressed pts suggest that it decline over time without significant difference with respect to the general population.

The novel adjuvanted recombinant zoster vaccine demonstrated lower humoral immune response in pts with B-NHL with respect to other pts, probably due to anti-CD20 therapy, while cellular immunity was not affected, although the small number of pts requires further investigation.

Very few data concerning persistence of immunity to childhood vaccines after anti-CD20-based therapy are available and suggest that humoral immunity to diphtheria and tetanus may be significantly impaired after therapy.

This is a prospective biological study evaluating the persistence of COVID-19 vaccine and other vaccines' (zoster, diphtheria and tetanus)-induced immunity in a subgroup of FL patients undergoing frontline induction immuno-chemotherapy and anti-CD20 maintenance within the prospective FIL_FOLL19 study (NCT05058404).

After the signature of a specific informed consent, eligible patients will receive a questionnaire evaluating vaccination history, past infection history and treatment, and passive immune prophylaxis (e.g. tixagevimab/cilgavimab administration). A baseline blood sample will be collected before the initiation of treatment and will be sent to the central laboratory, where specific analyses evaluating vaccine-induced cellular and/or humoral immunity against COVID-19, VZV, diphtheria and tetanus will be performed.

COVID-19 cellular and humoral immunity will be evaluated in all patients at all available timepoints.

Humoral and cellular immunity for VZV will be evaluated for all patients at study entry. In the subgroup of patients with a detectable serologic response at study entry, humoral and cellular immunity will be also evaluated at all available later timepoints.

Humoral immunity for diphtheria and tetanus will be evaluated for all patients at study entry. In the subgroup of patients with a detectable serologic response at study entry, humoral immunity will be also evaluated at all available later timepoints.

T-cell immunological parameters will be evaluated at study entry and 12 months after EOI (or early withdrawal).

ELIGIBILITY:
Inclusion Criteria:

1. Enrolment in FIL_FOLL19 study
2. Previous vaccination for COVID-19 (at least 3 doses)
3. Availability of informations about COVID-19 and other vaccines previously administered (vaccination records)
4. Willingness to comply with blood collection timepoints required for vaccination immunity evaluation
5. Signature of specific informed consent form

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Follicular Lymphoma undergoing frontline induction immuno-chemotherapy and anti-CD20 maintenance within the prospective FIL_FOLL19 study
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with persistence of cell-mediated immunity induced by COVID-19 approved vaccines (at least three doses) after standard induction immuno-chemotherapy. | At the end of induction therapy (EOI) - About 8 months from treatment start
  Proportion of patients with laboratory parameters of vaccine-induced cellular immunity against SARS-CoV-2 (by ELISpot assay) at EOI (after induction immuno-chemotherapy) vs proportion at baseline

SECONDARY OUTCOMES:
Rate of patients with persistence of cell-mediated immunity induced by COVID-19 approved vaccines (at least three doses) during anti-CD20 mAbs maintenance | At +12 months of maintenance - About 20 months from treatment start
  Proportion of patients with laboratory parameters of vaccine-induced cellular immunity against SARS-CoV-2 (by ELISpot assay) during anti-CD20 maintenance (+12 months after EOI) vs proportion at baseline
Rate of patients with persistence of humoral immunity induced by COVID-19 approved vaccines (at least three doses) after standard induction immuno-chemotherapy and during maintenance. | At the end of induction therapy (EOI) and at +12 months of maintenance - About 8 months and 20 months from treatment start respectively
  Proportion of patients with laboratory parameters of vaccine-induced humoral immunity against SARS-CoV-2 (by ELISA assay detecting anti-receptor binding domain [RBD] and anti-nucleocapsid [N] IgG antibodies) after standard induction immuno-chemotherapy (EOI) and during anti-CD20 maintenance (+12 months after EOI) vs proportion at baseline (excluding patients who received pre-exposure tixagevimab/cilgavimab or other monoclonal antibodies).
Rate of patients (with a detectable serologic response at study entry) with persistence of humoral and cellular immunity induced by adjuvanted recombinant zoster vaccine after standard induction immuno-chemotherapy and during maintenance | At the end of induction therapy (EOI) and at +12 months of maintenance - About 8 months and 20 months from treatment start respectively
  Proportion of patients with laboratory parameters of vaccine-induced humoral (by ELISA assay detecting anti-glycoprotein E IgG antibodies) and/or cellular immunity (by ELISpot assay) against VZV at EOI and during anti-CD20 maintenance (+12 months after EOI) vs proportion at first detection after vaccination (in the subgroup of patients with a detectable serologic response at study entry).
Rate of patients (with a detectable serologic response at study entry) with persistence of humoral immunity induced by childhood vaccines (diphtheria and tetanus) after standard induction immuno-chemotherapy and during maintenance | At the end of induction therapy (EOI) and at +12 months of maintenance - About 8 months and 20 months from treatment start respectively
  Proportion of patients with laboratory parameters of vaccine-induced humoral immunity against diphtheria and tetanus (by ELISA assay detecting diphtheria toxin-binding IgG and tetanus toxoid-binding IgG) at EOI and during anti-CD20 maintenance (+12 months after EOI) vs proportion at baseline (in the subgroup of patients with a detectable serologic response at study entry).
Rate of COVID-19 infection events and severity in vaccinated patients and correlation with humoral and/or cellular immunity with eventual tixagevimab/cilgavimab or other MAb prophylaxis and with dominant SARS-CoV-2 variant/subvariant at time of infection | From baseline (before therapy) up to 20 months from treatment start (+12 months of maintenance)
  Incidence of COVID-19 infections and their severity in vaccinated patients undergoing induction immuno-chemotherapy and maintenance and correlation with the level of immunity as measured by humoral and/or cellular immune parameters at the time point before the event as well as with eventual tixagevimab/cilgavimab administration (or prophylaxis with other monoclonal antibodies) and with dominant SARS-CoV-2 variant/subvariant at the time of infection
Rate of zoster infection events and their severity in vaccinated patients and correlation with the level of immunity as measured by humoral and/or cellular immune parameters at the time point before the event | From baseline (before therapy) up to 20 months from treatment start (+12 months of maintenance)
  Incidence of zoster infections and their severity in vaccinated patients undergoing induction immuno-chemotherapy and maintenance and correlation with the level of immunity as measured by humoral and/or cellular immune parameters at the time point before the event.
Characterization of multiple T-cell immunological parameters before and after standard induction immuno-chemotherapy in patients with follicular lymphoma treated within the prospective FIL_FOLL19 study | From baseline (before therapy) up to 20 months from treatment start (+12 months of maintenance)
  Description in the study population at study entry and at the latest timepoint of the percentage and absolute number of T lymphocytes populations and their subset distribution, expression of markers of activation and of functional exhaustion and immune checkpoints on T lymphocytes and T helper (Th) polarization of the CD4+ T-cell population by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Michele Merli, MD, Principal Investigator — U.O.C Ematologia, Ospedale di Circolo, Varese
Locations (14):
- Italy (14):
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino, AV
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, S.C. Ematologia, Alessandria, IT
  - Nuovo Ospedale degli Infermi, SSD Ematologia, Biella, IT
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan, IT
  - Ospedale Maggiore Policlinico Fondazione IRCCS Ca' Granda - Ematologia, Milan, IT
  - A.O.U. Maggiore della Carità di Novara - S.C.D.U. Ematologia, Novara, IT
  - IRCCS Policlinico San Matteo - Divisione di Ematologia, Pavia, IT
  - Ospedale Guglielmo da Saliceto - U.O. Ematologia, Piacenza, IT
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia U, Torino, IT
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia, Torino, IT
  - ASST Spedali Civili - S.C. Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - A.O.U. Senese - U.O.C. Ematologia, Siena